CLINICAL TRIAL: NCT01776827
Title: Long-term Outcome of Laparoscopic Hiatal Hernia Repair With or Without Alloderm Mesh at a University Hospital
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: LifeCell (Industry)
Responsible Party: Sponsor
Other Study IDs: 0168-12-FB
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia; Paraesophageal Hernia
Keywords: GERD; Hiatal Hernia; Paraesophageal Hernia; Biologic Mesh
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To study the long term outcome of Laparoscopic Hiatal Hernia Repair with human acellular dermal matrix Alloderm (LifeCell, Branchburg, NJ) mesh.

DETAILED DESCRIPTION:
To study the long term outcome of Laparoscopic Hiatal Hernia Repair with human acellular dermal matrix Alloderm (LifeCell, Branchburg, NJ) mesh. A barium swallow test with x-rays will be performed to look for recurrence of hiatal hernia. If the participants are symptomatic, additional medical therapy will be provided as deemed appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent paraesophageal hernia repair at UNMC.
* Greater than 19 years of age
* Not pregnant

Exclusion Criteria:

* Children and adolescents
* Pregnant and breast-feeding patients
* Vulnerable subjects such as decisionally impaired persons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent paraesophageal hernia repair at the University of Nebraska Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-05-22 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2015-02-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of hiatal hernia or GERD symptoms | 3+ years after initial surgery
  Patients will be questioned concerning their gastroesophageal reflux symptoms and hernia recurrence will be assessed using a barium swallow and x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Oleynikov, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States